CLINICAL TRIAL: NCT02925351
Title: The Biodistribution of 18F-Clofarabine in Patients With Autoimmune and Inflammatory Diseases
Brief Title: Fluorine F 18 Clofarabine PET/CT in Imaging Patients With Autoimmune or Inflammatory Diseases
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-001600; NCI-2016-01303 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-001600 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2016-09-08; First posted 2016-10-05 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2019-11

CONDITIONS: Autoimmune Disease; Crohn Disease; Inflammatory Disorder; Rheumatoid Arthritis; Systemic Lupus Erythematosus; Takayasu Arteritis
MeSH Terms: conditions — Autoimmune Diseases; Crohn Disease; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Takayasu Arteritis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imaging (fluorine F 18 clofarabine, PET/CT) (Experimental): Patients receive fluorine F 18 clofarabine IV and undergo a single PET/CT scan for up to 120 minutes.
  Interventions: Procedure: Computed Tomography; Radiation: Fluorine F 18 Clofarabine; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Radiation: Fluorine F 18 Clofarabine — Given IV
  Other Names: 18F-CA; 18F-Clofarabine; [18F]-Clofarabine; Cl-18F-ara-A
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot trial studies how well fluorine F 18 clofarabine positron emission tomography (PET)/computed tomography (CT) works in imaging patients with autoimmune or inflammatory diseases. Fluorine F 18 clofarabine is an imaging agent or tracer which may be taken up by inflammatory tissue in the body. Diagnostic imaging, such as PET/CT scans, can be used to measure the amount of injected tracer that is taken up by inflammatory tissue. PET/CT scan may help to determine how fluorine F 18 clofarabine is distributed throughout the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine how fluorine F 18 clofarabine (18F-clofarabine) is distributed in the body, in patients with autoimmune and inflammatory diseases.

II. Determine whether 18F-clofarabine can be used to image patients with autoimmune and inflammatory diseases.

OUTLINE:

Patients receive fluorine F 18 clofarabine intravenously (IV) and undergo a single PET/CT scan for up to 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older.
* Diagnosed with an autoimmune and inflammatory disorder.

Exclusion Criteria

* Women of childbearing age will have to undergo a pregnancy test that will be provided free of charge.
* Patients unable to undergo or comply with PET/CT scanning due to pre-existing medical conditions including claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Standardized Uptake Value | Baseline up to 240 minutes after injection
  Standardized Uptake Value (SUV) will be the primary unit for assessment. Using standard PET/CT viewing software, the SUV will be measured for different organs and lesions of suspected disease and compared to reference/background tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Allen-Auerbach, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States